CLINICAL TRIAL: NCT00230126
Title: A Phase II Randomized Study of OSI-774 in African American Patients With Advanced and Previously Treated Non-Small Cell Lung Cancer (NSCLC)
Brief Title: OSI-774 in African American Patients With Advanced and Previously Treated Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0443; NCI-2011-03221 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: African Americans
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A erlotinib 150 mg (Active Comparator): erlotinib 150 mg/day cycles 1 - 3
  Interventions: Drug: erlotinib
- B erlotinib modified according to weight (Experimental): erlotinib Cycle 1 dose modified according to patient's weight; Cycles 2 and up, dose titrated to skin rash.
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
  Other Names: Tarceva

SUMMARY:
This study determines tumor response rate, time to tumor progression and survival rate at 1 year produced by OSI-774 in previously treated African American patients with nonsmall cell lung cancer.

DETAILED DESCRIPTION:
Rationale: Researchers are seeking to identify treatment regimens with low toxicity for non-small cell lung cancer (NSCLC), especially for African Americans with this disease who seem to have a larger burden of comorbidities and decreased performance status. The current study uses a drug called OSI-774 in previously treated African American patients with NSCLC. OSI-774 is a targeted agent designed as an EGFR tyrosine kinase inhibitor. Previous research indicates that tumor cells overexpress EGFR receptors, and this drug works by blocking these receptors on tumor cells that that help them grow.

OSI-774 is FDA approved for the treatment of patients with non-small cell lung cancer that had been previously treated with chemotherapy. Unfortunately, very little data exist in the pharmacokinetics and metabolism of EGFR blockers in African Americans and in the assessment of how efficacious these agents are in this patient group. Yet, research suggests that EGFR blockage may have a greater impact on this patient population. Since the development of skin rash following therapy with EGFR blockers may be a surrogate of obtaining sufficient concentrations at the tissue level and potential efficacy, the current study is a randomized phase II trial designed to compare normal dose levels of OSI-774 with dose levels determined by body weight and with subsequent amounts adjusted further into the study to generate a skin rash. Through the current study, researchers are testing their theory that this dosing method will increase the number of patients with effective tissue concentrations and result in an increase in patient responses.

Purpose: The primary objective of this study is to determine the objective tumor response rate, the time to tumor progression, and the survival rate at one year produced by OSI-774 in previously treated African American patients with advanced NSCLC. A second objective is to evaluate if a regimen of single agent OSI-774, with dosing initially influenced by body weight and with subsequent titration to achieve skin rash is a suitable regimen for future studies of this agent. A third objective is to measure if changes in EGFR from tumor and blood cells correlate with the development of rash and clinical benefit. The pharmacokinetics of OSI-774 will also be characterized through study participants.

Treatment: Patients in this study will be given OSI-774. A computer will randomly assign patients into one of two treatment groups. Group one will be given a standard dose of OSI-774. The dose of OSI-774 will not be increased in group one. However, patients in group one will have the dose level decreased due to unacceptable side effects. Group two will receive OSI-774 at a dose modified to their body weight at study entry and subsequently adjusted further into the study to generate a skin rash. For all study participants, OSI-774 will be administered daily in oral pills. Several tests and exams will be given throughout the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed stage IIIB or IV NSCLC treated with 1-2 platinum- or taxane-containing regimens
* Measurable disease
* May have had prior surgery & external beam radiation
* African American
* 18 years or older

Exclusion Criteria:

* Known brain mets
* Prior treatment with EGFR targeting therapies
* Pregnant/lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2005-10; Primary Completion 2011-09 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villalona, M.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Erlotinib 150 mg/Day: 150 mg/day cycles 1 - 3
  erlotinib: Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
- Arm B: Erlotinib 150 to 200 mg/Day Depending on Body Weight; C: Cycle 1 dose modified according to patient's weight; Cycles 2 and up, dose titrated to generate skin rash.
  erlotinib: Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
Period: Overall Study
Arm/Group | Arm A: Erlotinib 150 mg/Day | Arm B: Erlotinib 150 to 200 mg/Day Depending on Body Weight; C
Started | 30 | 28
Completed | 28 | 27
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Fifty-eight patients . 31 men, 24 women.
Groups:
- Arm A: 150 mg/Day: 150 mg/day
  erlotinib: Arm A: 150 mg/day Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
- Arm B: Cycle 1 - 150-200 mg/Day Depending on Body Weight: Cycle 1 dose modified according to patient's weight; Cycles 2 and up, dose titrated to generate skin rash.
  Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
- Total: Total of all reporting groups
Arm/Group | Arm A: 150 mg/Day | Arm B: Cycle 1 - 150-200 mg/Day Depending on Body Weight | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Median (Full Range); unit: years] | 63 [29 to 83] | 59 [37 to 96] | 62 [29 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate at 12 Weeks
Description: no progression of disease at 12 weeks from starting treatment
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Erlotinib: Arm A: 150 mg/Day Cycles 1 - 3.: 150 mg/day cycles 1 - 3
  erlotinib: Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
- Arm B: Cycle 1 - 175 or 200 mg/Day Depending on Body Weight; C: Cycle 1 dose modified according to patient's weight; Cycles 2 and up, dose titrated to generate skin rash.
  erlotinib: Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
Arm/Group | Erlotinib: Arm A: 150 mg/Day Cycles 1 - 3. | Arm B: Cycle 1 - 175 or 200 mg/Day Depending on Body Weight; C
Number analyzed (Participants) | 26 | 26
participants | 6 | 6

2. Primary Outcome: Time to Progression
Time Frame: Every 12 weeks
Measure: Median (95% Confidence Interval); unit: months
Groups:
- A Erlotinib 150 mg/Day Cycles 1 - 3: erlotinib 150 mg/day cycles 1 - 3
  erlotinib: Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
- B Erlotinib Cycle 1 Dose Modified According to Weight: erlotinib Cycle 1 dose modified according to patient's weight; Cycles 2 and up, dose titrated to skin rash.
  erlotinib: Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
Arm/Group | A Erlotinib 150 mg/Day Cycles 1 - 3 | B Erlotinib Cycle 1 Dose Modified According to Weight
Number analyzed (Participants) | 26 | 26
months | 2.8 [2.5 to 3.1] | 2.4 [1.5 to 2.7]

3. Primary Outcome: 1-year Survival Rate
Time Frame: 12 months
Measure: Number; unit: percentage of patients
Arm/Group | A Erlotinib 150 mg/Day Cycles 1 - 3 | B Erlotinib Cycle 1 Dose Modified According to Weight
Number analyzed (Participants) | 26 | 26
percentage of patients | 30 | 26

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Arm A: 150 mg/Day Cycles 1 - 3: 150 mg/day cycles 1 - 3
  erlotinib: Arm A: 150 mg/day cycles 1 - 3. Arm B: Cycle 1 - 175 or 200 mg/day depending on body weight; Cycle 2 - if rash developed, then 150 mg/day; if no rash, then 175 mg/day; Cycle 3 - if rash developed, then 175 mg/day; if no rash, then 200 mg/day.
Arm/Group | Arm A: 150 mg/Day Cycles 1 - 3 | Arm B: Cycle 1 - 175 or 200 mg/Day Depending on Body Weight; C
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/27
Other Adverse Events (participants affected / at risk) | 19/28 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 150 mg/Day Cycles 1 - 3 (N=28) | Arm B: Cycle 1 - 175 or 200 mg/Day Depending on Body Weight; C (N=27)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: 150 mg/Day Cycles 1 - 3 (N=28) | Arm B: Cycle 1 - 175 or 200 mg/Day Depending on Body Weight; C (N=27)
rash (Skin and subcutaneous tissue disorders) | 19 | 19
Nausea/vomitting (Gastrointestinal disorders) | 2 | 6
diarrhea (Gastrointestinal disorders) | 9 | 7
anorexia (Gastrointestinal disorders) | 9 | 7 — not severe

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less